CLINICAL TRIAL: NCT03449888
Title: Arm Exercise Versus Pharmacologic Stress Testing for Clinical Outcome Prediction
Brief Title: Arm Exercise Versus Pharmacologic Stress Testing for Clinical Outcome
Acronym: ArmCrank
Status: Terminated | Type: Observational
Why Stopped: Terminated by the local IRB
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA St. Louis Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CARA-008-17F; 1 101 CX001345-01A3 (Other: VA St. Louis Health Care System)
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Veterans Referred to the St. Louis VAMC Stress Tes
MeSH Terms: interventions — regadenoson

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- St. Louis VA Healthcare System stress testing referrals: St. Louis VA Healthcare System cardiac stress testing laboratory referrals who are eligible and willing to complete an arm exercise ECG stress test, a treadmill ECG stress test if able, a regadenoson myocardial perfusion imaging stress test, and a coronary artery calcium score and cardiac computed tomographic angiography evaluation within 60 days if not referred for invasive coronary arteriography.
  Interventions: Procedure: Regadenoson myocardial perfusion imaging stress test; Procedure: Arm exercise electrocardiographic stress test; Procedure: Treadmill electrocardiographic stress test; Procedure: Coronary artery calcium score and cardiac computed tomographic angiography

INTERVENTIONS:
Procedure: Regadenoson myocardial perfusion imaging stress test — Best fit model of pharmacologic myocardial perfusion imaging data, including summed stress and difference scores, gated left ventricular ejection fraction, transient ischemic dilatation, and heart rate response to regadenoson data.
  Other Names: Lexiscan
Procedure: Arm exercise electrocardiographic stress test — Published arm exercise score and best fit model of arm exercise ECG stress testing data.
  Other Names: Arm exercise ECG
Procedure: Treadmill electrocardiographic stress test — Duke Treadmill Score and best fit model of treadmill exercise ECG stress testing data.
  Other Names: Treadmill ECG
Procedure: Coronary artery calcium score and cardiac computed tomographic angiography — Coronary artery calcium score by Agatston criteria and severe obstructive coronary artery disease > 70% by cardiac computed tomographic angiography or invasive coronary arteriography.
  Other Names: Coronary calcium score and cardiac CTA

SUMMARY:
This is a 5-year clinical trial to evaluate whether arm exercise electrocardiographic (ECG) stress testing without or with coronary artery calcium scoring (-/+ CAC) is non-inferior to treadmill ECG stress testing -/+ CAC and pharmacologic myocardial perfusion imaging as an initial evaluation to detect obstructive coronary artery disease, determined by cardiac computed tomographic angiography (CTA) and to predict clinical outcome, defined by a primary clinical endpoint of the composite of cardiovascular (CV) mortality, myocardial infarction, and 90-day post-stress test coronary artery revascularization and secondary clinical endpoints of all-cause mortality and CV mortality.

DETAILED DESCRIPTION:
Note: Recruitment is temporarily suspended because of VA-ORD moratorium due to Covid-19 pandemic. 04/01/2020

Treadmill exercise capacity and other physiologic responses to leg exercise are powerful predictors of mortality and provide important clinical and diagnostic information. However, many Veterans cannot perform treadmill exercise because of lower extremity or other disabilities. For many years, pharmacologic myocardial perfusion imaging (MPI) has been the standard of care for their evaluation but fails to provide powerful prognostic and clinically relevant information of exercise testing, requires exposure to ionizing radiation, and is several times more expensive than exercise electrocardiography (ECG). With a recently completed Merit Review award, we obtained substantial retrospective observational evidence that arm exercise ECG stress testing scores are at least equivalent to pharmacologic MPI for robust prediction of mortality and other measures of clinical outcome in Veterans who cannot perform leg exercise. Major hypotheses for the current proposal are: 1) arm exercise ECG stress testing scores or best fit models without or with coronary artery calcium scoring (-/+ CACS) are non-inferior to the Duke Treadmill Score -/+ CACS, best fit model treadmill ECG and regadenoson (r) MPI stress testing, all performed in the same Veterans in randomized order, as an initial evaluation for obstructive coronary artery disease (oCAD), and 2) arm exercise ECG stress testing scores or best fit models -/+ CACS are non-inferior to the Duke Treadmill Score -/+ CACS, best fit model treadmill ECG and rMPI stress testing in the same Veterans for predicting the primary clinical endpoint (composite of cardiovascular (CV) mortality, myocardial infarction, or 90-day post-stress test coronary revascularization) and secondary clinical endpoints of all-cause mortality and CV mortality. Our specific aim for all Veterans referred to the St. Louis Veterans Administration (VA) stress testing laboratory and are without exclusions for exercise or regadenoson stress testing or cardiac computed tomographic angiography (CTA), is to perform a single site prospective clinical trial comparing arm exercise ECG stress test scores and best models -/+ CACS with the Duke Treadmill Score -/+ CACS if able to perform treadmill exercise, and best fit treadmill ECG and rMPI models, all performed in the same Veterans, for identification of the diagnostic endpoint of oCAD, defined as a severely ( 70%) occluded epicardial, graft, or 50% left main coronary artery lumen, determined by cardiac CTA or invasive coronary arteriography, and prediction of the primary and secondary clinical endpoints described above. The arm exercise scoring system to be evaluated incorporates the variables arm exercise capacity in resting metabolic equivalents, 1-minute heart rate recovery and arm exercise-induced ST depression of 1 mm or greater. Regadenoson MPI variables to be evaluated include an abnormal MPI study and best fit models of summed stress and difference scores, transient ischemic dilatation, gated left ventricular ejection fraction, and the heart rate response. We plan to enroll 75 Veterans per year for 4 years and follow the entire cohort for an additional year. Statistical analyses will be performed with SAS using univariate and multivariate logistic and Cox regression models. We will evaluate non-inferiority of arm exercise scores -/+ CACS for their association with oCAD and prediction of clinical endpoints with a non-inferiority margin of 0.05. A long term goal is to develop a multi-site prospective randomized VA Cooperative Study to assess generalizability of arm exercise ECG stress testing -/+ CACS for diagnostic and prognostic evaluation in the VA and United States healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Any veteran referred to the St. Louis VA Healthcare System stress testing laboratory for a cardiac stress test

Exclusion Criteria:

* Contra-indications to stress testing such as acute coronary syndrome, uncompensated heart failure, or unstable cardiac dysrhythmias Inability to perform arm exercise stress testing
* Contra-indications to regadenoson stress testing such as significant reversible airway disease, heart block, or low blood pressure
* An abnormal baseline ECG (e.g. left bundle branch block, widespread ST segment depression of at least 1 mm, ventricular paced rhythm) that precludes interpretation of the stress ECG
* Contra-indications to cardiac computed tomographic angiography (CTA) such as contrast allergies and renal dysfunction (glomerular filtration rate < 30 ml/min)

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any veteran referred to the St. Louis VA Healthcare System stress testing laboratory
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Composite of cardiovascular mortality, myocardial infarction, and 90-day post-stress test coronary artery revascularization | 5 years
  Death from a cardiovascular cause, occurrence of myocardial infarction, and 90-day post-stress test coronary artery revascularization by any technique determined from VA, National Death Index, Missouri Health and Human Services, and non-VA medical records, and patient follow-up information.

SECONDARY OUTCOMES:
All-cause mortality | 5 years
  Death from any cause determined from VA, Social Security, and National Death Index records and patient follow-up information.
Cardiovascular mortality | 5 years
  Death from a cardiovascular cause determined from VA, Missouri Health and Human Services, and National Death Index records and patient follow-up information.

OTHER OUTCOMES:
Obstructive coronary artery disease | 5 years
  Severely (at least 70%) or completely occluded epicardial coronary arteries or grafts determined by cardiac computed tomographic angiography or invasive coronary arteriography

CONTACTS AND LOCATIONS:
Overall Officials: Wade H. Martin, MD, Principal Investigator — St. Louis VA Medical Center John Cochran Division, St. Louis, MO
Locations (1):
- St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available indefinitely after completion of the study 6/30/2023
Access Criteria: Data will be made available to outside investigators for purposes approved by the Principal Investigator, Co-investigators and St. Louis VA Healthcare System Institutional Review Board